CLINICAL TRIAL: NCT00251511
Title: A Phase II Trial of Trisenox Plus Thalomid as Treatment in Patients With Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor terminated trial
Sponsor: Veeda Oncology (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-04-001
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Arsenic Trioxide

SUMMARY:
This is a Phase II, open-label, non-randomized study in patients with low, intermediate-1, intermediate-2, or high-risk MDS (defined by IPSS).

Each cycle of treatment will be 6 weeks in length. Patients will be evaluated every 6 weeks for response. Patients will be treated for a minimum of 12 weeks even in the absence of response. Following 12 weeks of treatment, patients will continue to receive study treatment until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the study, patients must fulfill all of the following criteria:

  1. Patients must have signed an IRB-approved informed consent.
  2. Patients with low, intermediate-1, intermediate-2, and high-risk MDS (defined by IPSS) with documented diagnosis of MDS (refractory anemia, refractory anemia with excess blasts, refractory anemia with ringed sideroblasts, refractory anemia with mixed lineage dysplasia, or chronic myelomonocytic leukemia).
  3. Patients must have a documented history of all transfusions (pRBC and/or platelets) received in the 60-day period prior to their initial Trisenox treatment on this protocol.
  4. Patients with ECOG Performance Status of 0 or 1 (see Appendix I).
  5. Absolute QT interval below 460 msec in the presence of serum potassium and magnesium values within the normal range.
  6. Patients must be >/= 18 years of age.
  7. Patients must either be not of child bearing potential or have a negative serum pregnancy test within 24 hours prior to registration. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or they are postmenopausal for at least 24 months.
  8. For patients of childbearing potential, patient has agreed to use 2 reliable forms of contraception simultaneously for at least 1 month before beginning Thalomid therapy, during Thalomid therapy, and for 1 month following discontinuation of Thalomid therapy.
  9. Renal function: creatinine < 1.5 x institutional upper limit of normal (ULN), CTCAE Grade 1.
  10. Hepatic function: bilirubin </= 1.5 x ULN, CTCAE Grade 1. AST </= 2.5 x ULN, CTCAE Grade 1.
  11. Serum potassium >4.0mEq/dL and serum magnesium >1.8 mg/dL.

Exclusion Criteria:

* Any of the following criteria will make the patient ineligible to participate in this study:

  1. Patients who have received prior chemotherapy or prior therapy with either Trisenox or Thalomid.
  2. Patients who have a history of hypersensitivity to arsenic or thalidomide or any of the components in these drugs.
  3. Patients with a significant history of cardiac disease (i.e., uncontrolled hypertension, unstable angina, congestive heart failure, or myocardial infarction in the last 6 months).
  4. Patients with a history of torsade de pointes.
  5. Patients planning to receive any concurrent therapy to treat MDS during the study treatment period.
  6. Patients with a serious uncontrolled intercurrent medical or psychiatric illness, including serious infection.
  7. Patients with a history of other malignancy within the last 5 years, which could affect the diagnosis or assessment of these study drugs for MDS.
  8. Any patient who is pregnant or lactating.
  9. Any patient who is unable to comply with requirements of study.
  10. Patients with peripheral neuropathy >grade 1.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-08; Primary Completion 2006-01 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Primary Study Endpoint:
Determine the response rate (by IWG criteria) of patients with low, intermediate-1, intermediate-2, or high-risk MDS (defined by IPSS) to biweekly Trisenox plus daily Thalomid

SECONDARY OUTCOMES:
Secondary Study Endpoint(s):
Determine the toxicities associated with a biweekly Trisenox plus daily Thalomid regimen, the event-free survival, and the overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Boccia, MD, Principal Investigator — Veeda Oncology
Locations (1):
- Veeda Oncology, Houston, Texas, United States